CLINICAL TRIAL: NCT05979844
Title: MDMA-assisted Brief Cognitive Behavioral Conjoint Therapy for PTSD
Acronym: MDMA-bCBCT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Leslie Morland (U.S. Federal Agency)
Collaborators: Healing Breakthrough (Unknown); Lykos Therapeutics (Industry); San Diego Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Dr. Leslie Morland, Dr. Leslie Morland, San Diego Veterans Healthcare System
Organization: San Diego Veterans Healthcare System (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IVAPT2
Record Dates: First submitted 2023-07-31; First posted 2023-08-07 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: PTSD; Relational Problems
Keywords: PTSD; Intimate relationships; MDMA
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: An open label, single site study assessing the preliminary effectiveness, safety, and acceptability of an intervention consisting of MDMA-assisted bCBCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Non-medicine sessions of bCBCT + Medicine Sessions with 3,4-methylenedioxymethamphetamine (MDMA) (Experimental): bCBCT Non-medicine sessions: 8 sessions
  MDMA Medicine sessions:
  Initial Dose 1: 80 mg MDMA HCl (~68 mg MDMA) Supplementary Dose 1: 40 mg MDMA HCl (~34 mg MDMA) Initial Dose 2: 100 mg MDMA HCl (~84 mg MDMA) Supplementary Dose 2: 40 mg MDMA HCl (~34 mg MDMA)
  Interventions: Drug: 3,4-methylenedioxymethamphetamine (MDMA); Behavioral: Brief Cognitive Behavioral Conjoint Therapy (bCBCT)

INTERVENTIONS:
Drug: 3,4-methylenedioxymethamphetamine (MDMA) — 2 MDMA sessions; PTSD+ Veteran partner only
Behavioral: Brief Cognitive Behavioral Conjoint Therapy (bCBCT) — 8 bCBCT sessions; Both partners

SUMMARY:
The goal of this pilot trial is to examine the preliminary effectiveness of MDMA-facilitated bCBCT for improving chronic PTSD and relationship functioning in a sample of veterans and their intimate partners seeking care within the VA San Diego Healthcare System.

DETAILED DESCRIPTION:
The pilot study is a single site, open-label study assessing the preliminary effectiveness, safety, and acceptability of MDMA-assisted therapy in combination with brief Cognitive Behavioral Conjoint Therapy in a sample of 8 veterans diagnosed with PTSD and their intimate partners (N = 16) within the Veterans Affairs San Diego Healthcare System (VASDHS). Therapy teams will deliver the 8 session bCBCT intervention combined with two full-day MDMA sessions for the Veteran diagnosed with PTSD. The veteran with PTSD will be given 80 mg of MDMA HCl with a 40 mg MDMA HCl supplemental dose in the first session and 100 mg of MDMA HCl with a supplemental dose of 40 mg MDMA HCl in the second. The intimate partner will be present for the MDMA sessions (unless they decline or it is clinically contraindicated) but will not receive MDMA. The couples will complete one preparatory session and at least two Emotion Focused Integrative sessions (five max). The PTSD+ veteran will receive telephone check-in calls every other business day for one week following each MDMA session. The first MDMA session occurs in the morning the business day after the preparatory session and the second MDMA session occurs in the morning within 5 business days after bCBCT Session 7. The Emotion-Focused Integrative Sessions take place the morning after each MDMA session. Outcomes examining PTSD symptom severity and relationship functioning will be evaluated for preliminary effectiveness. The study's screening, enrollment, and baseline phase lasts from pre-screen to baseline (approximately 12 weeks, +/- 2 weeks). The treatment period lasts from bCBCT Session 1 to bCBCT Session 8 (7 weeks -13 weeks). The follow-up period lasts from the post-treatment assessment to study termination (24 weeks +/- 15 days).

ELIGIBILITY:
Inclusion Criteria:

1. Be a veteran (age 18 years or older) who meets criteria for PTSD on the CAPS-5 or be an intimate partner (age 18 or older) of a veteran meeting the criteria for PTSD who is willing to participate in the intervention and who does not meet criteria for PTSD on the PCL-5 (i.e., must score a 30 or lower).
2. Be in a committed relationship together of at least 12 months, and be cohabiting.
3. Be fluent in speaking and reading English.
4. Are willing to commit to medication dosing, therapy sessions, follow-up sessions, completing evaluation instruments, and all necessary telephone contact.
5. Be able to swallow pills. (PTSD+ veteran only)
6. Agree to have study visits recorded, including Experimental MDMA Sessions, and be aware that Independent Rater assessments for bCBCT sessions will occur.
7. Provide a contact (relative, spouse, close friend, or other support person) who is willing and able to be reached by the investigators in the event of a participant becoming suicidal or unreachable. (PTSD+ veteran only)
8. Agree to inform the investigators within 48 hours of any new medical conditions or procedures.
9. If able to become pregnant (i.e., assigned female at birth, fertile, following menarche and until becoming post-menopausal unless permanently sterile), must have a highly sensitive negative pregnancy test at study entry and prior to each Experimental MDMA Session, and must agree to use adequate birth control through 10 days after the last Experimental MDMA Session. Adequate birth control methods include intrauterine device (IUD), injected, implanted, intravaginal, or transdermal hormonal methods, abstinence, oral hormones plus a barrier contraception, vasectomized sole partner, or double barrier contraception. Two forms of contraception are required with any barrier method or oral hormones (i.e., condom plus diaphragm, condom or diaphragm plus spermicide, oral hormonal contraceptives plus spermicide or condom). (PTSD+ veteran only)
10. Agree to the following lifestyle modifications: comply with requirements for fasting and refraining from certain medications prior to Experimental MDMA Sessions. (PTSD+ veteran only)
11. Not enroll in any other interventional clinical trials during the duration of the study, and commit to medication dosing, therapy, and study procedures.
12. Both partners agree to not begin a new form of mental healthcare during the screening or treatment phases of the trial, without first discussing with the PI in consultation with the study physician.

    1. It is acceptable for participants to continue ongoing non-PTSD focused or non-couple-based mental healthcare, if it is not increased in frequency or specifically excluded by the study protocol.
    2. All ongoing therapies should be documented by the site and discussed with the study physician prior to enrollment to avoid confounding treatment effects. In some instances, the study physician may request that the participant delay enrollment until their planned course of therapy is complete, and an integration period has elapsed.
    3. Participants may continue with PTSD focused and/or couple-based mental health care during the screening period prior to Baseline and following treatment period prior to study termination if they have approval from the study PI and their study provider (as applicable).

    Medical History - PTSD+ veteran only unless otherwise noted
13. At Pre-Screening, have at least moderate PTSD symptoms in the last month based on PCL-5 total score of 40 or greater (index).
14. May have well-controlled hypertension that has been successfully treated with anti- hypertensive medicines if they pass additional screening to rule out underlying cardiovascular disease.
15. May have asymptomatic Hepatitis C virus (HCV) that has previously undergone evaluation and treatment as needed.
16. At Screening, have at least moderate PTSD per CAPS-5 and symptoms in the last month constituting a CAPS-5 Total Severity Score of 28 or greater (index).
17. May have alcohol or substance use disorder if participant is not in withdrawal or requiring detox. Participants/couples must have a plan, agreed upon by investigator, therapy team, and study physician, to reduce use of alcohol or other substances and to manage symptoms without self-medicating. Enrollment will require that, in the judgment of the investigator, therapy team, and study physician, the plan for decreasing substance use is realistic and has a good chance of succeeding in order to prevent substance use from impacting the safety or effectiveness of the investigational treatment. (Both partners)
18. May have a history of or current Diabetes Mellitus (Type 2) if additional screening measures rule out underlying cardiovascular disease, if the condition is judged to be stable on effective management, and with approval by the study physician.
19. May have hypothyroidism if taking adequate and stable thyroid replacement medication.
20. May have a history of, or current, glaucoma if approval for study participation is received from an ophthalmologist.

Exclusion Criteria:

1. Are not able to give adequate informed consent.
2. Are currently engaged in compensation and pension (C&P) litigation whereby financial gain would be achieved from prolonged symptoms of PTSD or any other psychiatric disorders.
3. Are likely, in the investigator's opinion and via assessment period, to be re- exposed to their index trauma or other significant trauma, lack social support, or lack a stable living situation
4. Have used Ecstasy (material represented as containing MDMA) more than 10 times within the last 10 years or at least once within 6 months of the first Experimental MDMA Session. (PTSD+ veteran only)
5. Have any current problem which, in the opinion of the investigator or study physician, might interfere with participation due to it impacting the patient's safety and/or ability to participate in the protocol
6. Have hypersensitivity to any ingredient of the Investigational Medicinal Product (IMP). (PTSD+ veteran only)

   Psychiatric History - both members of dyad unless otherwise noted
7. Have received Electroconvulsive Therapy (ECT) within 12 weeks of enrollment. (PTSD+ veteran only)
8. Have a history of or a current primary psychotic disorder assessed via the DIAMOND and clinical interview
9. Have a history of or a current Bipolar I disorder, Bipolar 2 disorder, or manic episode assessed via the DIAMOND and clinical interview (PTSD+ veteran only)
10. Have a current eating disorder with active purging assessed via DIAMOND and clinical interview. (PTSD+ veteran only)
11. Have current major depressive disorder with psychotic features assessed via DIAMOND
12. Have current panic disorder assessed via DIAMOND (PTSD+ veteran only)
13. Have a current alcohol or substance use disorder other than caffeine or nicotine that the investigators, therapy team, and/or study physician judge to be a safety concern for enrollment in the study or that could interfere with the therapeutic process or with other aspects of study participation. Any participant who is not able to agree or adhere to a plan to reduce use and manage symptoms will not be enrolled
14. Present with current serious suicide risk, as determined through psychiatric interview, responses to C-SSRS (scores of four or greater), and clinical judgment of the investigator; however, history of suicide attempts is not an exclusion. Any participant who is likely to require hospitalization related to suicidal ideation and behavior, in the judgment of the investigator, will not be enrolled. Any participant presenting with the following on the pre-screen C-SSRS will be excluded:

    1. Suicidal ideation score of 4 or greater within the last 6 months of the assessment at a frequency of once a week or more
    2. Any suicidal behavior, including suicide attempts or preparatory acts, within the last 6 months of the assessment. Participants with non-suicidal self- injurious behavior may be included if approved by the study physician
15. Report intimate partner violence or severe relationship aggression, as defined by meeting either of the following criteria, that that the investigators and/or therapy team judge to be a safety concern for enrollment in the study or that could interfere with the therapeutic process or with other aspects of study participation:

    1. A score of ≥7 on the Extended - Hurt, Insult, Threaten, Scream (E-HITS) screening tool
    2. A score of "severe" on the Psychological Aggression scale of the Revised Conflict Tactics Inventory (CTS-2)
16. Would present a serious risk to others as established through clinical interview and if necessary, discussion with treating psychiatrist
17. Require ongoing concomitant therapy with a psychiatric medication other than the exceptions described in protocol section on Concomitant Therapy. (PTSD+ veteran)

    Medical History - PTSD+ veteran only
18. Have a history of any medical condition that could make receiving a sympathomimetic drug harmful because of increases in blood pressure and heart rate. This includes, but is not limited to, a history of myocardial infarction, cerebrovascular accident, or aneurysm. Participants with other mild, stable chronic medical problems may be enrolled if the study physician and PI agree the condition would not significantly increase the risk of MDMA administration or be likely to produce significant symptoms during the study that could interfere with study participation or be confused with side effects of the IMP. Examples of stable medical conditions that could be allowed include, but are not limited to Diabetes Mellitus (Type 2), Human Immunodeficiency Virus (HIV) infection, Gastroesophageal Reflux Disease (GERD), etc. Any medical disorder judged by the investigator to significantly increase the risk of MDMA administration by any mechanism would require exclusion.
19. Have a diagnosis of uncontrolled hypertension defined by the American Heart Association as repeated readings of ≥ 140 millimeters of Mercury [mmHg] systolic or ≥ 90 mmHg diastolic
20. Have a history of ventricular arrhythmia at any time, other than occasional premature ventricular contractions (PVCs) in the absence of ischemic heart disease
21. Have Wolff-Parkinson-White syndrome or any other accessory pathway that has not been successfully eliminated by ablation
22. Have a history of arrhythmia, other than premature atrial contractions (PACs) or occasional PVCs in the absence of ischemic heart disease, within 12 months of screening. Participants with a history of atrial fibrillation, atrial tachycardia, atrial flutter or paroxysmal supraventricular tachycardia or any other arrhythmia associated with a bypass tract may be enrolled only if they have been successfully treated with ablation and have not had recurrent arrhythmia for at least one year off all antiarrhythmic drugs and confirmed by a cardiologist
23. Have a marked Baseline prolongation of QT/QTc interval. For purposes of eligibility, this is defined as repeated demonstration of a QT interval corrected using Fridericia's formula [QTcF] >450 milliseconds [ms]
24. Have a history of additional risk factors for Torsade de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
25. Require use of concomitant medications that prolong the QT/QTc interval during Sessions. Refer to protocol section on Concomitant Medications
26. Have symptomatic liver disease or have significant liver enzyme elevations
27. Have history of hyponatremia or hyperthermia
28. Weigh less than 48 kilograms (kg)
29. Are pregnant or nursing or are able to become pregnant and are not able/willing to practice an effective means of birth control
30. Have engaged in ketamine-assisted therapy or used ketamine within 12 weeks of enrollment
31. Have any preexisting conditions that can affect renal functioning

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-10-06 (Actual); Primary Completion 2025-11-14 (Actual); Study Completion 2025-11-14 (Actual)

PRIMARY OUTCOMES:
Clinician-rated PTSD symptoms | Baseline - 6 months post-treatment
  Measured using the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5). The CAPS-5 is a 20-item diagnostic interview that asks about the severity of four PTSD-related symptom clusters: re-experiencing, avoidance, negative alterations in cognition and mood, and alterations in arousal and reactivity. The evaluator rates responses on a 5-point Likert scale (0 = Absent to 4 = Extreme/Incapacitating). Total scores range from 0 to 80 with higher scores indicating greater severity.

SECONDARY OUTCOMES:
Relationship satisfaction | Baseline - 6 months post-treatment
  Measured using the Couples Satisfaction Index (CSI-32). The CSI-32 is a 32-item self-report survey that measures romantic relationship satisfaction. The first item measures the overall happiness of the relationship on a 7-point scale (0 = Extremely unhappy to 6 = Perfect). The other 31 items capture satisfaction, quality, and happiness of the relationship on 6-point scales (0 to 5) with varying response options. Total CSI-32 scores range from 0 to 161 with higher scores indicating greater relationship satisfaction. Scores below 104.5 indicate clinical relationship distress.

OTHER OUTCOMES:
Suicidality | Baseline - 6 months post-treatment
  Measured using the Columbia Suicide Severity Rating Scale (C-SSRS). The C-SSRS is designed to assess suicidal ideation, ideation intensity, and behaviors during a clinical trial.
Self-reported PTSD symptoms | Baseline - 6 months post-treatment
  Measured using the PTSD Checklist for DSM-5 (PCL-5). The PCL-5 is a 20 item self report questionnaire that asks about the presence and severity of PTSD symptoms. The participant rates their distress caused by PTSD symptoms on a 5-point Likert scale (1 = Not at all to 5 = Extremely). Total scores range from 0-80, with higher scores indicating greater severity. Partners will complete the collateral version of the PCL-5 (PCL-C) starting at Baseline.
Emotion regulation | Baseline - 6 months post-treatment
  Measured using the Emotional Regulation Questionnaire (ERQ). The ERQ is a 10-item self-report questionnaire that asks about the use of cognitive reappraisal and expressive suppression to alter emotion. Participants respond using a 7-point Likert scale (1= Strongly disagree to 7=Strongly agree). Higher scores indicate higher use of cognitive reappraisal and/or expressive suppression.
Adverse childhood events | Baseline
  Measured using the Adverse Childhood Events Scale (ACES). The ACES is a 10-item self-report survey that asks about childhood stress. Participants indicate exposure to different kinds of abuse with yes/no responses, and answer with "1" if the abuse happened often. Higher scores indicate greater exposure to childhood stressors.
Relationship conflict | Baseline - 6 months post-treatment
  Measured using the Short Form of the Revised Conflict Tactics Scale (CTS-2S). The CTS-2S is a self-report inventory with 10 paired items that asks about conflict and intimate partner violence across 5 domains. The participant evaluates their own actions and the partner's actions for each of the 10 items, making 20 items total. Participants respond using an ordinal scale from 0 (This has never happened) to 6 (More than 20x in the past year).
Depressive symptoms | Baseline - 6 months post-treatment
  Measured using the Beck Depression Inventory II (BDI-II). The BDI-II is a 21-item self-report measure that asks about depression symptom severity. Participants rate the severity of each symptom on a scale of 0 to 3. Total scores range from 0-63, with higher scores indicating higher severity.
Sleep | Baseline - 6 months post-treatment
  Measured using the Pittsburgh Sleep Quality Index (PSQI). The PSQI is a 19-item self-report questionnaire that asks about 7 subcategories of sleep quality over the last month. Participants respond using a combination of Likert scales (from 0 to 3) and open-ended questions that are later converted to scaled scores. Higher total scores indicate greater sleep disturbance.
Trauma exposure | Baseline
  Measured using the Life Events Checklist for DSM-5 (LEC-5). The LEC-5 is a 17-item self-report survey that asks about exposure to potentially traumatic events. Participants check off the type of exposure for each event (Happened to me, Witnessed it, Learned about it, Part of my job, Not sure, Doesn't apply).
Posttraumatic growth | Baseline - 6 months post-treatment
  Measured using the Posttraumatic Growth Inventory (PTGI). The PTGI is a 21-item self-report measure that asks about level of posttraumatic growth across 5 subscales in adults who have experienced trauma. Participants respond using a 6-point Likert scale (1=I did not experience this change as a result of my crisis, to 6=I experienced this change to a very great degree as a result of my crisis).Total scores range from 1-126.
Symptom accommodation | Baseline - 6 months post-treatment
  Measured using the Significant Others' Response to Trauma Scale (SORTS). The SORTS is a 28-item self-report measure of a partner's accommodating behaviors for a patient's PTSD symptoms. Participants rate the frequency and intensity of 14 accommodating behaviors using a scale of 0-4. Higher scores indicate greater accommodation.
Satisfaction with care | Post-Assessment (~1 week after intervention)
  Measured using the 8-item version of the Client Satisfaction Questionnaire (CSQ-8). The CSQ-8 asks about patient satisfaction with healthcare and services they received. Participants respond using a Likert scale from 0-3 with varying response options for each question. Higher scores indicate higher satisfaction.
Treatment expectations | Baseline
  Measured using the Stanford Expectations of Treatment Scale (SETS). The SETS is a 10-item self-report questionnaire that assesses a patient's feelings about their upcoming treatment. The first 6 items are rated on a 7-point Likert scale (1=strongly disagree, to 7=strongly agree). Items 7-9 are open-ended. Item 10 is a yes/no response. The scale yields a score for positive expectancy and negative expectancy.
Sexual Functioning | Baseline - 6 months post-treatment
  Measured using the Changes in Sexual Functioning Questionnaire (CSFQ-14). The CSFQ-14 is a 14-item self-report scale that evaluates sexual functioning. The five subscales are: pleasure, desire/frequency, desire/interest, arousal/excitement, and orgasm/completion. All items are scored on 5-point scales with varying response options. Higher total scores indicate better sexual functioning. The CSFQ-14 has corresponding assigned-male-at-birth and assigned-female-at-birth versions.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Morland, Principal Investigator — San Diego Veterans Healthcare System
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Morland LA, Perivoliotis D, Wachsman TR, Alam A, Knopp K, Khalifian C, Ramanathan D, Chargin BE, Bismark AW, Glynn S, Stauffer C, Wagner AC. MDMA-assisted brief cognitive behavioral conjoint therapy for PTSD: Study protocol for a pilot study. Contemp Clin Trials Commun. 2024 May 24;40:101314. doi: 10.1016/j.conctc.2024.101314. eCollection 2024 Aug. PMID 38994348